CLINICAL TRIAL: NCT05525286
Title: A Multicentric Phase 1/2 Trial to Evaluate the Safety and Efficacy of SOT102 as Monotherapy and in Combination With Standard of Care Treatment in Patients With Gastric and Pancreatic Adenocarcinoma
Brief Title: Clinical Trial of SOT102 Antibody Drug Conjugate in Patients With Advanced Gastric and Pancreatic Adenocarcinoma
Acronym: CLAUDIO-01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Trial terminated by Sponsor based on benefit- risk reassessment
Sponsor: SOTIO Biotech a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SN201; 2021-005873-25 (EudraCT Number); 2023-504441-31-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-07; First posted 2022-09-01 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: SN201 is a multi-modular clinical trial in patients with pancreatic adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg (Experimental): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.032 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
  Interventions: Drug: SOT102
- SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg (Experimental): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.064 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
  Interventions: Drug: SOT102
- SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg (Experimental): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.128 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
  Interventions: Drug: SOT102
- SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg (Experimental): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.214 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
  Interventions: Drug: SOT102
- SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg (Experimental): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.,32 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes. Upon completion of the SOT102 infusion, first-line SoC treatment was administered. SoC treatment was nab-paclitaxel (125 mg/m2) given as a 30- to 40-minute infusion followed by gemcitabine (1000 mg/m2) given as a 30-minute infusion on days 1, 8, and 15. This treatment was repeated every 28 days.
  Interventions: Drug: SOT102

INTERVENTIONS:
Drug: SOT102 — SOT102 is an antibody-drug conjugate (ADC) targeting CLDN18.2 with the anthracycline PNU as cytotoxic moiety.

SUMMARY:
This trial will assess the MTD and RP2D of SOT102 administered as monotherapy (Part A) and in combination with first-line SoC treatment (nab-paclitaxel/ gemcitabine; Part B) and efficacy of SOT102 administered as monotherapy (Part C) and in combination with first-line SoC treatment (Part D) in patients with advanced or metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
The trial will have the following parts:

* Part A: Dose escalation, first-in-human, single-agent phase 1 trial of SOT102 in advanced/metastatic pancreatic cancer patients with unmet medical need (CLDN18.2 agnostic)
* Part B : Phase 1b dose escalation combination trial of SOT102 in combination with nab-paclitaxel/gemcitabine as SoC regimen for first-line treatment of patients with advanced/metastatic pancreatic cancer (CLDN18.2 agnostic)

Once an RP2D in the respective phase 1 evaluation (Part A and Part B) has been identified, expansion parts (Part C and Part D) are planned:

* Part C : Single-agent SOT102 expansion at RP2D identified in Part A in pancreatic cancer after one or more prior systemic therapies (second+ line) for locally advanced or metastatic disease (CLDN18.2 positive)
* Part D : SOT102 in combination with nab- paclitaxel/gemcitabine for first-line treatment expansion at RP2D identified in Part B in pancreatic cancer (CLDN18.2 positive)

ELIGIBILITY:
Inclusion Criteria:

All Parts (key criteria)

* Hematologic: Absolute neutrophil count ≥1.5×10⁹/L, platelets ≥100×10⁹/L, hemoglobin ≥9 g/dL
* Hepatic: Bilirubin ≤1.5× upper limits of normal (ULN), ALT and AST ≤2.5×ULN; in case of liver involvement: AST and ALT ≤5×ULN
* Renal: Creatinine clearance ≥60 mL/min calculated by Cockcroft-Gault formula
* Prothrombin time/international normalized ratio (INR) ≤1.5×ULN
* Albumin ≥3.0 mg/dL
* Proteinuria <1 g/24 hours
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Estimated life expectancy ≥3 months as per investigator's assessment
* A female patient is eligible to participate if she is not pregnant, not breastfeeding, not of childbearing potential/ agreed with contraception

Part A

* Patient has advanced inoperable or metastatic disease
* Patient has no better treatment option available
* Measurable or non-measurable disease according to RECIST 1.1
* Histological or cytological evidence of adenocarcinoma of pancreas that is advanced or metastatic

Part B (in addition to relevant A criteria)*Histological or cytological evidence of adenocarcinoma of the pancreas that is advanced or metastatic (pancreas)

Part C (in addition to relevant A criteria)*Must have received at least one prior systemic therapy for advanced or metastatic disease (pancreas)

Part D (in addition to relevant B criteria)*Histological or cytological evidence of adenocarcinoma of the pancreas that is advanced inoperable or metastatic (pancreas)

Exclusion Criteria:

All Parts (key criteria)

* Patient has received radiation therapy ≤14 days before day 1 of cycle 1 or has not recovered to grade ≤1 from treatment-related side effects
* Severe preexisting medical conditions as per judgement of the investigator (e.g., active gastric or GEJ ulcer with or without bleeding, complete or incomplete gastric outlet syndrome with persistent or repetitive bleeding)
* History of interstitial pneumonitis or pulmonary fibrosis
* Symptomatic central nervous system malignancy. Patients with asymptomatic or treated central nervous system metastases may be eligible if they are not treated with corticosteroids or anticonvulsants and the disease is stable for at least 60 days.
* Patient has peripheral sensory neuropathy grade ≥2
* Active infection requiring systemic therapy within ≤7 days prior to day 1 of cycle 1
* History of major ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, Torsades de Pointes)
* Bradycardia (<50 beats per minute)
* Family history of sudden cardiac death before age 50
* History or family history of congenital long QT syndrome
* Major surgical intervention ≤28 days prior to ICF signature or incomplete wound healing after surgical intervention
* Time since last transfusion of RBCs ≤14 days before cycle 1 day 1
* Vaccination with a live or live-attenuated vaccine within 30 days prior the first dose of trial interventions

Part B/D (key)

*Patients with contraindications to any component of the first-line SoC treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, M.D., Ph.D., Principal Investigator — Vall d'Hebron University Hospital (HUVH)
Locations (8):
- United States (2):
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Cleveland Clinic Main Campus, Cleveland, Ohio
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
- Masarykův Onkologický Ústav, Brno, Czechia
- Institut Gustave Roussy, Paris, France
- Spain (2):
  - VHIO - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Dose Level 1: 0.032 mg/kg
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Started | 4 | 0 | 0 | 0 | 4
Completed | 4 | 0 | 0 | 0 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2: 0.064 mg/kg
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Started | 0 | 11 | 0 | 0 | 0
Completed | 0 | 11 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3: 0.128 mg/kg
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Started | 0 | 0 | 9 | 0 | 0
Completed | 0 | 0 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4: 0.214 mg/kg
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SOT102 as Monotherapy (Part A) DL2 0.046 mg/kg: Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.064 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
- SOT102 in Combination With SoC (Part B) 0.032 mg/kg: Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with 0.032 mg/kg of SOT102 given once every 14 days via the IV route over 45 (±15) minutes. Upon completion of the SOT102 infusion, first-line SoC treatment was administered. SoC treatment was nab-paclitaxel (125 mg/m2) given as a 30- to 40-minute infusion followed by gemcitabine (1000 mg/m2) given as a 30-minute infusion on days 1, 8, and 15. This treatment was repeated every 28 days.
- Total: Total of all reporting groups
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.046 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) 0.032 mg/kg | Total
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 10 | 6 | 1 | 4 | 24
  >=65 years | 1 | 1 | 3 | 2 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (6.95) | 55.4 (9.62) | 57.6 (9.67) | 65.3 (2.08) | 51.8 (2.63) | 56.5 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 2 | 2 | 12
  Male | 3 | 8 | 5 | 1 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 7 | 1 | 4 | 23
  Unknown or Not Reported | 0 | 4 | 2 | 2 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 7 | 7 | 1 | 4 | 23
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 2 | 2 | 0 | 8
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 3 | 3 | 1 | 1 | 8
  Czechia | 2 | 0 | 3 | 0 | 3 | 8
  United States | 0 | 3 | 0 | 0 | 0 | 3
  France | 0 | 3 | 1 | 1 | 0 | 5
  Spain | 2 | 2 | 2 | 1 | 0 | 7
ECOG status [Count of Participants; unit: Participants] — As per the Inclusion criteria, only patients with ECOG performance status ≤1 (i.e., ECOG performance status 0 or 1) could participate in the trial. This measure shows distribution of the status across safety population. As per the ECOG status scale, 0 means patients who are fully active, able to carry on all pre-disease performance without restriction. 1 means patients, who are restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Participants
    0 | 2 | 4 | 3 | 2 | 2 | 13
    1 | 2 | 7 | 6 | 1 | 2 | 18
Weight at baseline [Mean (Standard Deviation); unit: kilograms] | 77.8 (16.58) | 75.5 (22.3) | 72.7 (18.08) | 62.7 (21.02) | 72.4 (19.54) | 73.4 (19.08)
Height at baseline [Mean (Standard Deviation); unit: meters] | 1.74 (0.12) | 1.74 (0.135) | 1.73 (0.107) | 1.67 (0.195) | 1.69 (0.101) | 1.72 (0.121)
BSA at baseline [Mean (Standard Deviation); unit: square meters] | 1.90 (0.271) | 1.89 (0.311) | 1.86 (0.288) | 1.67 (0.379) | 1.83 (0.263) | 1.86 (0.287)

OUTCOME MEASURES:

1. Primary Outcome: Parts A and B: The Definition of the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of SOT102 Given as Monotherapy and in Combination With First-line SoC Treatment
Description: MTD is defined as the highest dose level tested below the dose level associated with ≥33% of dose-limiting toxicity (DLT)-evaluable patients experiencing a DLT. The RP2D will be selected based on evaluation of the totality of all data. The trial was halted early due to safety signals not initially deemed DLTs that were seen across different dose levels. After a protocol amendment formally defined this signal as a DLT, the trial was restarted, but the same safety signal reappeared. Following a review by the independent Dose Escalation Committee, the trial was terminated.
Time Frame: Through Cycles 1-2 (28 days)
Population: DLT evaluable patients were those who have received 2 doses of SOT102 per schedule (day 1 of cycle 1 and day 1 of cycle 2) with the maximum postponement of cycle 2 by 1 day (as agreed by the sponsor) and completed the evaluation period of 28 days. Also patients who experienced a treatment emergent adverse event at any time during the DLT evaluation period that met the definition of a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- SOT102 as Monotherapy (Part A): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with escalating doses of SOT102 given once every 14 days via the IV route over 45 (±15) minutes.
- SOT102 in Combination With SoC (Part B): Patients with CLDN18.2-positive pancreatic adenocarcinoma were treated with escalating doses of SOT102 given once every 14 days via the IV route over 45 (±15) minutes. Upon completion of the SOT102 infusion, first-line SoC treatment was administered. SoC treatment was nab-paclitaxel (125 mg/m2) given as a 30- to 40-minute infusion followed by gemcitabine (1000 mg/m2) given as a 30-minute infusion on days 1, 8, and 15. This treatment was repeated every 28 days.
Arm/Group | SOT102 as Monotherapy (Part A) | SOT102 in Combination With SoC (Part B)
Number analyzed (Participants) | 20 | 1
Participants | NA — The protocol-defined MTD was never reached, since ≥33% of patients never had a DLT at any given dose level | NA — The protocol-defined MTD was never reached, since ≥33% of patients never had a DLT at any given dose level

2. Primary Outcome: Parts C and D: The Assessment of the Efficacy of SOT102 in Monotherapy and in Combination With First-line SoC Treatment
Description: Efficacy is determined by objective response rate (ORR) determined according to RECIST 1.1 criteria
Time Frame: From Day 1 of Cycle 1 until disease progression or start of new anticancer therapy, whichever is first, to be assessed up to approximately 4 years
Population: Part C and Part D were not initiated, no population was analyzed.
Groups:
- SOT102 in Monotherapy or in Combination With SoC - Expansion Cohorts: Patients were to be treated with SOT102 at the RP2D identified in Part B either as a monotherapy given once every 14 days via the IV route over 45 (±15) minutes or in combination with SoC. Upon completion of the SOT102 infusion, first-line SoC treatment was to be administered. SoC treatment was to be nab-paclitaxel (125 mg/m2) given as a 30- to 40-minute infusion followed by gemcitabine(1000 mg/m2) given as a 30-minute infusion on days 1, 8, and 15. This treatment was to be repeated every 28 days.
Arm/Group | SOT102 in Monotherapy or in Combination With SoC - Expansion Cohorts
Number analyzed (Participants) | 0

3. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With DLTs
Description: Adverse events (AEs) graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 considered DLTs: All grade 5 events not clearly related to disease progression or any other causes; Any grade 3 or higher non-hematologic toxicity regardless of duration; Grade 2 or higher serum creatinine elevation; Hy's law cases; Any grade 2 pneumonitis that does not resolve to grade 1 within 3 days of the initiation of maximal supportive care; Recurrent grade 2 pneumonitis; Grade 2 or higher proteinuria; Grade 4 neutropenia lasting more than 7 days; Febrile neutropenia; Grade 3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia. AEs NOT considered DLTs: Grade 3 nausea, vomiting, or diarrhea that can be controlled within 72 hours; Grade 3 fatigue less than 5 days; Grade 3 or higher correctable electrolyte abnormalities that last less than 72 hours and not associated with clinical complications; Grade 3 or higher amylase or lipase
Time Frame: Through Cycles 1-2 (28 days)
Population: Patients who received 2 doses of SOT102 per schedule (day 1 of cycle 1 and day 1 of cycle 2). Patients must have completed evaluation period of 28 days. Pancreatic patients must have received three doses of SoC (days 1, 8, and 15 of cycle 1), gastric patients must have received 2 doses of SoC per schedule (day 1 of cycle 1 and day 1 of cycle 2). Patients who experienced an adverse event at any time during the DLT evaluation period that met the definition of a DLT were included.
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 3 | 8 | 6 | 3 | 1
Participants | 0 | 1 | 1 | 0 | 0

4. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With Treatment-emergent AEs (TEAEs)
Description: A TEAE is defined as an AE that:
  * emerges during SOT102 treatment, having been absent at the time of pre-treatment (screening), or
  * re-emerges during SOT102 treatment, having been present at the time of pre-treatment (screening), or
  * worsens in severity during SOT102 treatment relative to the pre-treatment state if the AE is continuous.
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 4 | 10 | 9 | 3 | 4

5. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With SOT102-related AEs
Description: Causal relationship (relatedness) of all AEs will be assessed by investigators and classified as follows:
  * Not suspected: It is not plausible that the AE is caused by medication/procedure and a likely alternative explanation exists. No reasonable possibility of a causal or temporal relationship.
  * Suspected: It is plausible that the AE is caused by medication/procedure. Reasonable possibility of a causal relationship.
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.046 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 3 | 4 | 6 | 2 | 2

6. Secondary Outcome: Part B (Combination With SoC): Number of Participants With SoC-related AEs
Description: as for outcome 5
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SoC
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
Participants |  |  |  |  | 4

7. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With Serious AEs (SAEs)
Description: An SAE is any untoward medical occurrence that at any dose fulfills one or more of the following criteria:
  * Results in death
  * Is immediately life-threatening
  * Results in persistent or significant disability/incapacity Is a congenital anomaly/birth defect
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Is another medically significant event defined as an event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent any of the above listed outcomes
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 4 | 5 | 5 | 2 | 0

8. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With AEs Leading to Premature Discontinuation of SOT102
Description: AEs (intercurrent illness or trial treatment-related toxicity) that would, in the judgment of the investigator, affect assessments of clinical status to a significant degree or require discontinuation of trial treatment
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 0 | 1 | 3 | 1 | 0

9. Secondary Outcome: Part B (Combination With SoC): Number of Participants With AEs Leading to Premature Discontinuation of SoC
Description: as for outcome 8
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SoC
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4
Participants |  |  |  |  | 1

10. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants Who Died
Description: Date of death and immediate and underlying causes of death will be collected.
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 2 | 5 | 3 | 1 | 0

11. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With Clinical Laboratory Test Abnormalities (Coagulation, Hematology, Clinical Chemistry and Urinalysis) of Grade 3 or Higher Graded According to NCI CTCAE Version 5.0
Description: The following laboratory parameters will be assessed:
  * Coagulation: prothrombin time, INR
  * Hematology: leukocytes, erythrocytes, hemoglobin, hematocrit, platelets, differential
  * Clinical chemistry: ALT, albumin, ALP, amylase, AST, bilirubin, blood urea nitrogen or blood urea, calcium, creatinine, glucose (fasting), LDH, lipase, magnesium, potassium, sodium, TSH (gastric adenocarcinoma only)
  * Urinalysis: blood, glucose, ketones, pH, protein, specific gravity, urine leukocyte esterase
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 3 | 2 | 3 | 0 | 1

12. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Characterization of Cmax of SOT102
Description: Assessment of concentration of SOT102 and its derivates at various timepoints
Time Frame: From Day 1 of Cycle 1 until Day 1 of Cycle 5
Population: Patients who had at least 1 post-dose concentration measurement above the lower limit of quantification. No data was collected for Part B due to the low number of patients.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 10 | 9 | 3 | 0
ng/mL | 564.1750 [278.990 to 839.600] | 1220.3250 [853.400 to 2308.800] | 2792.6000 [281.060 to 3630.400] | 4980.6000 [3304.200 to 6304.000] |

13. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Characterization of Tmax of SOT102
Description: Assessment of concentration of SOT102 and its derivates at various timepoints
Time Frame: From Day 1 of Cycle 1 until Day 1 of Cycle 5
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 10 | 9 | 3 | 0
hours | 0.217 [0.17 to 3.02] | 0.217 [0.02 to 22.80] | 0.233 [0.02 to 3.13] | 0.233 [0.22 to 0.25] |

14. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Characterization of AUClast of SOT102
Description: Assessment of concentration of SOT102 and its derivates at various timepoints
Time Frame: From Day 1 of Cycle 1 until Day 1 of Cycle 5
Population: as for outcome 12
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 10 | 9 | 3 | 0
h*ng/mL | 44558.9495 [26130.047 to 72331.081] | 108104.0701 [37856.444 to 329008.958] | 321146.7316 [14143.478 to 458598.933] | 605136.8688 [461829.806 to 812024.200] |

15. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Evidence of SOT102 Activity in Monotherapy in Individual Patients - BOR: Complete Response
Description: Detection of anecdotal tumor response in individual patient, as per RECIST 1.1 criteria
Time Frame: From Day 1 of Cycle 1 until disease progression or start of new anticancer therapy, whichever is first, assessed up to approximately 2 years and 9 months
Population: Patients exposed to at least one dose of SOT102 who had at least one evaluable tumor assessment per RECIST v1.1 after the initiation of SOT102 treatment
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 2 | 9 | 8 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Evidence of SOT102 Activity in Monotherapy in Individual Patients - BOR: Partial Response
Description: Detection of anecdotal tumor response in individual patient, as per RECIST 1.1 criteria
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 2 | 9 | 8 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 1

17. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Evidence of SOT102 Activity in Monotherapy in Individual Patients - BOR: Stable Disease
Description: Detection of anecdotal tumor response in individual patient, as per RECIST 1.1 criteria
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 2 | 9 | 8 | 3 | 4
Participants | 1 | 3 | 2 | 1 | 3

18. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Evidence of SOT102 Activity in Monotherapy in Individual Patients - BOR: Progressive Disease
Description: Detection of anecdotal tumor response in individual patient, as per RECIST 1.1 criteria
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 2 | 9 | 8 | 3 | 4
Participants | 1 | 5 | 6 | 2 | 0

19. Secondary Outcome: Parts A and B (Monotherapy and Combination With SoC): Number of Participants With Antibodies Against SOT102
Description: Identification of patients who develop detectable antibodies against any part of SOT102
Time Frame: From Day 1 of Cycle 1 until 30 (+5) days after the last dose of SOT102, assessed up to approximately 2 years and 9 months
Population: Patients exposed to at least one dose of SOT102
Measure: Count of Participants; unit: Participants
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
Number analyzed (Participants) | 4 | 11 | 9 | 3 | 4
Participants | 3 | 2 | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to approximately 2 years and 8.5 months
Description: Only treatment-emergent adverse events were analyzed (see the definition above); the tables include information on treatment-emergent adverse events, serious treatment-emergent adverse events, and all deaths; causality was assessed by investigators
Arm/Group | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg
All-Cause Mortality (participants affected / at risk) | 2/4 | 5/11 | 3/9 | 1/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 4/4 | 5/11 | 5/9 | 2/3 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 9/11 | 8/9 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg (N=4) | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg (N=11) | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg (N=9) | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg (N=3) | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Protoeinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | NA
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Nephroangiosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOT102 as Monotherapy (Part A) DL1 0.032 mg/kg (N=4) | SOT102 as Monotherapy (Part A) DL2 0.064 mg/kg (N=11) | SOT102 as Monotherapy (Part A) DL3 0.128 mg/kg (N=9) | SOT102 as Monotherapy (Part A) DL4 0.214 mg/kg (N=3) | SOT102 in Combination With SoC (Part B) DL1 0.032 mg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (4)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (12)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 4 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (3)
Fatigue (General disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 4 (7)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (5)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Blood bilirubin increased (Hepatobiliary disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 4 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results will be published and/or presented at scientific meetings in their totality in a timely manner. Any formal publication of clinical trial results will be a collaborative effort between the sponsor and the investigator(s). All manuscripts or abstracts will be reviewed and approved in written by the sponsor before submission. The sponsor may request a delay in publication if there are important intellectual property concerns.

DOCUMENTS (2):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT05525286/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT05525286/SAP_002.pdf